CLINICAL TRIAL: NCT05294107
Title: Intestinal Organoids
Acronym: BIOÏDES
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 35RC21_8862_BIOÏDES
Record Dates: First submitted 2022-02-28; First posted 2022-03-24 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Digestive System Diseases; Inflammatory Bowel Disease, Ulcerative Colitis Type; Crohn Disease
Keywords: biobank; organoids; digestive disease; inflammatory bowel disease
MeSH Terms: conditions — Digestive System Diseases; Colitis, Ulcerative; Crohn Disease; Inflammatory Bowel Diseases

STUDY DESIGN:
Intervention Model Description: Prospective, monocentric cohort aiming at generating 3D organoids from human digestive samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group Crohn's disease (Experimental): 4 additional biopsies for 30 patients with Crohn's disease
  Interventions: Procedure: additional biopsies
- Group ulcerative colitis (Experimental): 4 additional biopsies for 30 patients with ulcerative colitis
  Interventions: Procedure: additional biopsies
- Group No MICI (Active Comparator): 4 additional biopsies for 30 patients out of Inflammatory Disease Chronic Bowel Disease
  Interventions: Procedure: additional biopsies

INTERVENTIONS:
Procedure: additional biopsies — After Verification of eligibility criteria, patient information and consent, digestive biopsies performed for the study are in addition to those performed for the patient's follow-up:
  * 6 biopsies are taken on average in clinical routine
  * 4 additional biopsies are necessary to obtain a sufficient number of amplifiable stem cells The samples will be sent within one hour to the Biological Resource Center of the University Hospital of Rennes at room temperature in a tube containing isotonic saline. (CRB).
  Biopsies will be then prepared by isolating intestinal crypts and cultured on a 3D matrix gel (matrigel) with added growth factors reproducing the niche environment of intestinal stem cells, which favors the development of an intestinal epithelium. After intestinal differentiation, organoids will be used for research such as molecular screening, assessment of the effects of intestinal stress and healing.

SUMMARY:
Over the last decade, the use of mini-organ or organoids has been increasingly developed in fundamental research. Indeed, digestive organoids represent an essential advance compared to classical culture systems (epithelial cell lines, immortalized cells) since they preserve in culture the functional complexity present in vivo (architecture, different cell types). They also have the advantage of being able to be propagated indefinitely (unlike explants), minimizing the use of animal models and reducing the amount of tissue required. Finally, their growth and development depends on the origin of the sample (the organoid will develop differently if the cell source comes from a patient suffering from an inflammatory bowel disease, for example), thus generating models of human pathologies to better determine their physiopathology. The use of organoids in biomedical research has proven to be an indispensable tool for the understanding of cellular and molecular mechanisms involved in epithelial renewal and the screening of molecules and ingredients for applications in the health and agri-food sectors.

DETAILED DESCRIPTION:
The project aims to generate a biocollection of 3D intestinal models from digestive biopsies with associated health data and to characterize them before using them for the screening of potential therapeutic molecules.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 18 to 75 years
* Subject undergoing endoscopy as part of the standard of care with the need to take digestive biopsy samples
* Subject having signed a free and informed consent in writing

Exclusion Criteria:

* Subjects under legal protection (safeguard of justice, curatorship or guardianship) or deprived of liberty.
* Anticoagulant treatment and anti-platelet treatment (except for aspirin 75 mg)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-09-06 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Number of isolated intestinal crypts per biopsies | Day 0
  Biopsies will be then prepared by isolating intestinal crypts and cultured on a 3D matrix gel (matrigel) with added growth factors reproducing the niche environment of intestinal stem cells, which favors the development of an intestinal epithelium. After intestinal differentiation, organoids will be used for research such as molecular screening, assessment of the effects of intestinal stress and healing.

SECONDARY OUTCOMES:
Number of differentiated organoids | Day 0
Fold change of MUC2 expression | Day 0
Fold change of LGR5 expression | Day 0
KI67 expression | Day 0

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume BOUGUEN, Professor, Principal Investigator — Rennes University Hospital
Locations (1):
- CHU de RENNES-Service des Maladies de l'Appareil Digestif, Rennes, France

IPD SHARING:
Plan to Share IPD: No